CLINICAL TRIAL: NCT03415880
Title: The Light Intensity Physical Activity Trial
Brief Title: Light Intensity Physical Activity Trial
Acronym: LiPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Principal Investigator, Annemarie Koster, PhD, Principal Investigator, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL57173.068.16
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus; Physical Exercise; Light Intensity Physical Activity; Arterial Stiffness; Aortic Stiffness; Pulse Wave Velocity; Type2 Diabetes; Sedentary Lifestyle; Artery Disease; Physical Activity
Keywords: Diabetes mellitus; Type2 Diabetes; Sedentary Lifestyle; Physical Activity; Pulse wave velocity; arterial stiffness; aortic stiffness; artery disease; light intensity physical activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The study consists of an intervention group and a control group. Both arms run parallel and both groups are measured at the same time points.
Who Masked: Investigator
Masking Description: The investigator measuring the outcome measures will be blinded to patient allocation. Patients are asked not to mention their allocated group or the programme they follow and not to wear or mention the wrist-worn activity tracker during measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Participants attend 4 workshops and undergo all measurements at t=0, t=3, t=6, and t=12 months.
  Interventions: Behavioral: Workshops control group LiPAT
- Intervention group (Experimental): Participants attend 4 workshops, receive a wrist-worn feedback physical activity monitor, a smartphone app, and telephone coaching. All participants undergo all measurements at t=0, t=3, t=6, and t=12 months.
  Interventions: Behavioral: Interactive workshops LiPAT intervention group; Device: Wrist-worn feedback physical activity monitor; Device: Smartphone application LiPAT; Behavioral: Telephone Coaching

INTERVENTIONS:
Behavioral: Interactive workshops LiPAT intervention group — Workshops include practical behavior change strategies and address barriers to movement, awareness of the immediate benefits of movement and implementation-intentions. Participants will be encouraged to cultivate a learning mind-set in order to better tolerate potential set-backs and to apply strategies such as pre-planning their week to incorporate physical activity, engaging their social network, and setting up systems and habits. Participants' progress in changing their physical activity patterns which will be compared and discussed.
  Arms: Intervention group
Device: Wrist-worn feedback physical activity monitor — Participants receive the feedback monitor (Fitbit inspire®; commercially available consumer product (https://www.fitbit.com/inspire)
  Arms: Intervention group
Device: Smartphone application LiPAT — With a cloud-based platform the iHealth data is synchronized with a mobile phone app developed by the research team. The app is designed to help the participant to self-monitor their physical activity levels and includes information on total activity and number of steps taken.
  Arms: Intervention group
Behavioral: Telephone Coaching — participants in the intervention group will receive telephone coaching during the first 3 months of the intervention. Telephone coaching will be conducted twice in the first month and once each in months two and three. The researcher will enquire about the progress with increasing LiPA, about the experiences of applying the strategies discussed during workshops, and about the experience with Fitbit Inspire® and the corresponding app. If needed, the coach will offer suggestions to improve goal adherence.
  Arms: Intervention group
Behavioral: Workshops control group LiPAT — During the first 6 months of the study (the intervention period) participants in the control group will attend 4 workshops in which the benefits of physical activity and the health-risks of sedentary behavior will be discussed. Additionally, information will be provided on healthy lifestyle for patients with type 2 diabetes.
  Arms: Control group

SUMMARY:
In type 2 diabetes (T2D), physical activity is an important modifiable risk factor of cardiovascular disease (CVD). Unfortunately (long-term) compliance to exercise programs in patients with T2D is poor. Light-intensity physical activity (LiPA) such as walking slowly, household activities or taking a flight of stairs might be a potential target for lowering the CVD risk in patients with T2D since it can perhaps be more be incorporated into daily life. To assess cardiovascular disease risk in this single-blinded RCT, the investigators settled on measuring arterial stiffness as the primary outcome. Arterial stiffness has independent predictive value for cardiovascular events and can be measured reliably and non-invasively. The investigators hypothesize that light intensity physical activity intervention program based upon increasing LiPA by replacing sedentary time is effective in lowering arterial stiffness as estimated by aortic pulse wave velocity (PWV) and carotid distensibility in individuals with T2D.

DETAILED DESCRIPTION:
Total duration of the RCT is 12 months, with the first 6 month as the intervention period and the last 6 months as follow-up.

Community-dwelling individuals with type 2 diabetes are eligible for participation in the trial, taking into account the in- and exclusion criteria described below, 160 participants will be included, 80 in each study arm. Study measurements of all participants will take place at baseline (month 1 (t = 0)), month 3 (t = 3), month 6 (t = 6, and month 12 (t = 12) at the Maastricht UMC+.

Participants in the intervention group will be instructed to increase their LiPA by decreasing sedentary time. Participants will follow 4 workshops in group sessions on strategies to change their physical activity behaviour and will receive a feedback physical activity monitor that will be worn continuously on the wrist and provide e-feedback on activity behaviour.

Participants in the control group will receive 4 workshops in group sessions on healthy lifestyle including information and strategies to increase LiPA and reduce sedentary time similar to the intervention group, but will not receive a feedback-activity monitor.

Screening A preliminary screening will be carried out by telephone interview. If eligibility criteria are met the participant will attend the baseline visit which starts with the informed consent procedure. Afterwards, a standard physical examination will take place and an ultrasound scan will be performed to screen for large atherosclerotic plaques of the carotid arteries. If the participant is indeed eligible for inclusion, the investigational baseline measurements are performed after which randomization will take place. From then on participants will run through the protocol either being part of the intervention or control group.

Measurements at the four investigational visits (t = 0, 3, 6 and 12)

* sociodemographic data
* medical history & medication use: by means of an interview
* lifestyle factors (alcohol use and smoking behaviour), quality of life, depressive symptoms - by means of questionnaires
* Sedentary and physical activity monitoring: by means of the activPAL® activity monitor for 7 days
* venous sampling (approx. 40 ml per person per visit; 8 collecting tubes of 5 ml) for fasting glucose, fasting insulin, HbA1c, lipid profile, creatinin, albumin and biomarkers of endothelial dysfunction (vWF, s-VCAM-1, sE-selectin, sTM, SICAM-1), low-grade inflammation(CRP, SAA, IL-6, TNF-alfa, IL-8) and immune cells. The remainder of the material will be stored in a biobank for future determination of any potentially interesting (bio)markers on the topic of physical activity. For any such future procedures further approval will be sought from the METC/MUMC+.
* Anthropometric data (height, weight, waist and hip circumference and bio-electrical impedance measurements)
* vascular measurement (arterial stiffness, microvascular function and blood pressure)
* physical function measurements (grip strength and timed chair test)
* Objective measurement of light-intensity physical activity through activPAL ® activity monitor that will be worn for 7 days continuously at baseline, month 3, month 6, and month 12. This device is blinded to the participant. Data from the activPAL provide detailed and accurate information on the participants' sedentary, standing, and stepping time for each day.

Sample size calculation In order to be able to detect a 10% difference in PWV and similarly a 10% difference in carotid distensibility (the primary objectives of the study) after the intervention between the intervention group and the control group, both groups should consist of at least 73 participants each if assuming a probability of a type 1 error at 0.05 (i.e., alfa) and an 80% (i.e., beta) ability to detect a true difference between the intervention group and the control group. These estimates are conservative taking into account only PWV values at entry and exit of the trial. The 10% difference is speculative and based upon a mean PWV estimates from 'The Maastricht Study' data as there is currently no data available on LiPA and arterial stiffness. In order to correct for potential drop out (roughly estimated at 10%) 80 participants will be included in each group.

Statistical analysis The significance levels used in the statistical analyses will be 0.05. The validity of the normality assumption will be check for all outcomes. Baseline characteristics will be compared between the intervention and the control group. For continuous variables (e.g. age, BMI) mean and standard deviations will be presented; numbers and percentages will be shown for categorical variables (e.g. smoking, medication use). T-tests will be used to compare differences in continuous baseline characteristics between the intervention and control group and chi-square test will be used for categorical variables. Assuming that the randomization was successful no differences are expected. Missing data will be imputed using multiple imputations techniques.

Primary study parameter(s) The effect of the intervention on the primary outcome PWV at month 6 will be analysed using intention-to-treat (ITT) approach according to randomization assignment. The ITT analyses will be used as primary method for our statistical analyses and any outcomes in our reports will be primarily based upon these ITT analyses. In addition, a per protocol analysis will be performed for those who attended the workshops. These analyses will be used to gain some insights into any potential non-response / drop out. These per protocol analyses will not be the primary source for reporting outcomes. General linear models will be used to analyse the effect of the intervention on PWV at month 6. Due to the COVID-19 crisis some month 6 measurement will take place at a later moment, depending on the duration of this delay we will have to adjust for this in our statistiscal anlayes. In addition, repeated measures will be taken into account, baseline, month 3, and month 6 using mixed models in SPSS. The 3-month visits might be missing for some particiapants due to COVID-19 crisis, we assume that the 6-month measurements for these particiaptns can take place as planned In these models, subject is entered as a random effect and intervention (categorical variable with 2 levels: 1: intervention; 2: control group) as a fixed effect .The baseline value of PVW and sex will be used as covariates in analyses.

Secondary study parameter(s) Sedentary time, as measured by the activPAL will be analysed as total sedentary minutes on an average day as well as the percentage of sedentary during wake time. Similarly, time standing and stepping, also derived from the activPAL data will be analysed. All metabolic health parameters and microcirculation measurements will also be analysed as continuous variables. Quality of life and mental functioning are also analysed as continuous variables. Finally, measures of body composition measures are also all continuous outcomes variables

Similar to the primary outcome analyses, general linear mixed models will be used the analyses the change the secondary outcome measures from baseline to month 6. Using mixed models, the repeated measures will be taken into account similar the analyses with the primary outcome.

All analyses, for the both primary and secondary outcomes will also be conducted for the follow-up (month 12 data) to examine the long-term effect of the intervention, taking into account all repeated measures (baseline, month 3, month 6) in a mixed model.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 years old
* having type 2 diabetes
* BMI 20-35 kg/m2
* having a sedentary lifestyle (i.e., self-reported moderate-to-vigorous physical activity < 150 minutes per week)
* willingness to undergo randomization
* being in the possession of personally owned smart phone

Exclusion Criteria:

* not being able to walk for 15 minutes for any (medical) reason
* currently engaged in an (medical) exercise program
* plan to move out of the study area in the next 12 months
* (digital) illiteracy or being unable to read Dutch
* a history of any cardiovascular event (including stroke) three months prior to possible inclusion
* a history of signs or symptoms of ischemic heart disease and(or) heart failure three months prior to possible inclusion
* a history or signs or symptoms of peripheral arterial disease three months prior to possible inclusion
* a history or signs or symptoms of severe diabetic neuropathy or diabetic foot ulcers three months prior to possible inclusion
* a history of sign or symptoms of severe diabetic retinopathy three months prior to possible inclusion
* a history or sign or symptoms of severe osteoarthritis or severe joint complaints three months prior to possible inclusion
* a history or signs or symptoms of COPD (eligible are those participants with a COPD Gold classification ≤ I)
* uncontrolled diabetes (i.e., uncontrolled hypo- or hyperglycaemia)
* uncontrolled hypertension (i.e., systolic / diastolic blood pressure ≥ 180 / 95 mmHg)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
The effect of a LiPA intervention program on reducing aortic carotid-to-femoral pulse-wave velocity (PWV) in patients with type 2 diabetes. | Change from baseline PWV at 6 months.
  Aortic (carotid to femoral) PWV will be determined by means of applanation tonometry. It will be calculated as the median of three consecutive PWV recordings.
The effect of a LiPA intervention program on increasing carotid distensibility in patients with type 2 diabetes. | Change from baseline carotid distensibility at 6 months.
  Carotid distensibility will be determined at the left common carotid by means of arterial ultrasound.

SECONDARY OUTCOMES:
Feasibility of a LiPA intervention program on reducing sedentary time as measured by activPAL | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Daily activity levels will be measured by activPAL3™ physical activity monitor. The participants will wear the device fixated on their upper leg for 8 consecutive days at each measurement moment. ActivPAL measures total standing time, sedentary time (sitting or lying down), and stepping time (physical activity).
The effect of a LiPA intervention on changes in blood pressure. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in blood pressure
The effect of a LiPA intervention on waist -circumference in cm. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in waist -circumference
The effect of a LiPA intervention on quality of life as measured through the Dutch versions of the EQ-5D questionnaire. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  The EQ-5D is a short questionnaire that covers five dimensions of health: Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety/Depression. The EQ-5D includes 5 questions with 5 answer options each, ranging from 1 ('no problems') to 5 ('severe limitation'). A summary index with a maximum score of 1 can be computed from these five dimensions by means of a converion table. A score of 1 indicates the best health status. Additionally, there is a visual analogue scale (VAS) to indicate the general health status with scores ranging from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine').
The effect of a LiPA intervention on depressive symptoms with the use a validated Dutch version of the 9-item Patient Health Questionnaire (PHQ-9). | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  The PHQ-9 is a self-administered questionnaire based on the DMS-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) criteria for a major depressive disorder. It comprises nine items rated on a 4-point scale, ranging from 0 = "not at all" to 3 = "nearly every day". The PHQ-9 scale will also be used as a dichotomous variable with a pre-defined cut-off level of 10, which represents the presence of clinically relevant depressive symptoms.
Feasibility of a LiPA intervention program on increasing standing and stepping time as measured by activPAL. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Daily activity levels will be measured by activPAL3™ physical activity monitor. The participants will wear the device fixated on their upper leg for 8 consecutive days at each measurement moment. ActivPAL measures total standing time, sedentary time (sitting or lying down), and stepping time (physical activity). Stepping time (physical activity) is further classified into higher intensity physical activity (minutes with a step frequency >110 steps/min during waking time) and lower intensity physical activity (minutes with a step frequency ≤110 steps/min during waking time).
The effect of a LiPA intervention on fasting blood glucose | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in fasting blood glucose.
The effect of a LiPA intervention on HbA1c. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in HbA1c.
The effect of a LiPA intervention on total cholesterol. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in total cholesterol.
The effect of a LiPA intervention on HDL- and LDL-cholesterol. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in HDL- and LDL-cholesterol.
The effect of a LiPA intervention on triglycerides. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in triglycerides
The effect of a LiPA intervention on glucose lowering medication. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in glucose lowering medication.
The effect of a LiPA intervention on hip -circumference in cm. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in hip -circumference
The effect of a LiPA intervention on body composition | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of any changes in body composition as measured by bio electrical impedance.
The effect of a LiPA intervention on quality of life as measured through the Dutch version of the SF-36 questionnaire. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  The SF-36 is a generic and easily self-administered quality of life instrument. The SF-36 questionnaire measures health on eight multi-item dimensions, covering functional status, well-being, and overall evaluation of health. In six of these eight dimensions, participants rate their responses on a three or six point scale. For each dimension, item scores are coded, summed, and transformed on to a scale from 0 (worst health) to 100 (best health).
The effect of a LiPA intervention program on immune cells. | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Measurement of circulating immune cells using flow cytometry from fresh whole blood. In addition, measurement of circulating cytokines to assess the activation state of immune cells, and store immune cells for functional tests.
The effect of a LiPA intervention program on microvascular function | Measured at baseline (t=0), after month 3 (t=3), month 6 (t=6) and 12 months after baseline (t=12).
  Microvascular function will be evaluated in both the retina and the skin. Which will be determined with the use of fundoscopy and Skin laser Doppler flowmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Coen D Stehouwer, MD, PhD, Principal Investigator — Academisch Ziekenhuis Maastricht; Annemarie Koster, PhD, Principal Investigator — Maastricht University; Ronald M Henry, MD, PhD, Principal Investigator — Academisch Ziekenhuis Maastricht
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will be able to share documents upon reasonable request and once the study results have been published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will be able to share documents upon reasonable request and once the study results have been published. The paper with study results is currently in preparation.
Access Criteria: Requests could be addressed to the PI's.

DOCUMENTS (1):
  • Study Protocol (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT03415880/Prot_001.pdf